CLINICAL TRIAL: NCT05162040
Title: PedaleoVR: Credibility, Usability and Intrinsic Motivation Study of a Virtual Reality Application for Lower Limb Motor Rehabilitation
Brief Title: PedaleoVR: Credibility, Usability and Intrinsic Motivation Study
Status: Completed | Type: Observational
Sponsor: Werium Assistive Solutions (Industry)
Collaborators: Centro Lescer (Unknown); Cajal Institute of the Spanish National Research Council (Other)
Responsible Party: Sponsor
Other Study IDs: UsabilityPedaleoVR
Record Dates: First submitted 2021-11-12; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Ataxia, Motor; Hemiparesis
MeSH Terms: conditions — Ataxia; Paresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental Group: Twenty participants joined the experimental group (15 males and 5 females, mean aged=61.10; SD=12.62) and provided written informed consent to be enrolled onto the study. Participants with neurological pathologies were diagnosed with (6) ischemic strokes, (1) hemorrhagic stroke, (1) thalamic stroke, (1) internal capsule stroke (3) traumatic brain injury (TBI), (1) Parkinson syndrome, (1) mixed axonal neuropathy with sensory demyelination, (1) progressive multifocal leukoencephalopathy, (1) secondary obstructive hydrocephalus, (1) angioma avernosus hemorrhage, (1) hemiprotuberancial hemorrhage - cavernoma, (1) ataxia and (1) cerebral artery aneurysm.
  Interventions: Device: Use of PedaleoVR

INTERVENTIONS:
Device: Use of PedaleoVR — All participants must undergo an evaluation of their motor skills through the application of physical assessment metrics performed by the physician. The metrics are the Timed Up-and-Go Test (TUG) and the 6-minute walk test.
  Next, they must perform a pedaling exercise on a bicycle or stationary pedaling station synchronizing the physical activity with the visual feedback from the virtual reality application. Two pedalling sets of 10 minutes each are performed, with 5 minutes of rest between sets. Finally, the participant is asked to rate the usability: System Usability Rating Scale (SUS), activity credibility (Credibility and Expectancy Questionnaire, CEQ) and intrinsic motivation (Intrinsic Motivation Inventory, IMI) of the virtual reality application.

SUMMARY:
The objective of this research is to combine the use of inertial systems with virtual reality in pedalling exercises in a pilot study with subjects with ataxia or hemiparesis. In particular, it is intended to evaluate the validity of the system as a physical training tool for pedalling exercises aimed at providing motivational visual stimuli and biofeedback based on pedalling cadence to improve the exercise experience and promote adherence to the subject's treatment.

Primary objectives:

* To study the estimation of pedalling cadence performed by the system/platform in subjects with hemiparesis or ataxia..
* To study the usability, credibility and intrinsic motivation characteristics of the platform

DETAILED DESCRIPTION:
The objective of this research is to evaluate patient adherence to pedalling-based exercise training using visual feedback and virtual reality pedalling cadence analysis. In addition, the usability, credibility and adherence promotion characteristics of the virtual reality platform will be studied.

Study phases:

The procedure will be carried out in the following phases detailed below:

Phase 1: Sample recruitment and participant information. Participants are recruited according to the inclusion and exclusion criteria. The subject is informed about the experimentation in which he/she is going to participate, its duration and the technical characteristics to be used in the study. characteristics to be used in the study. The data to be collected in the form of standardized questionnaires are explained to the subject. Personal data will not be collected. If the subject is suitable for participation, he/she will be asked to sign the corresponding informed consent form. Finally, 3 appointments with the patient will be arranged in accordance with the general schedule of the the general schedule of the experiment.

Phase 2: Familiarization practice with the instrumentation. These will be aimed at acquiring basic skills in the use of the synchronized use of the virtual reality environment synchronized with the pedalling task.

Phase 3: Experimentation and data acquisition.

A.1. Pre-assessment: The participant's motor skills are evaluated based on the application of physical assessment metrics by the physician. The metrics are the "Timed Up-and-Go" (TUG) test and the "6-minute walking" test. Participants with no visual defects, mild cognitive impairment and lower limb motor skills could be selected if they also meet the inclusion/exclusion criteria.

A.2. Validation session of the usability of the Virtual Reality Platform in patients with Ataxia or Hemiparesis. (Approx. 40 minutes) The intervention consists of a pedalling exercise performed on a bicycle or static pedalling station while synchronizing the physical activity with the visual feedback of the virtual reality application. Two pedalling sets of 10 minutes each are performed, with 5 minutes of rest between sets.

A.3. Objective Evaluation: Once the exercise task of the first session is completed, the participant is asked to rate its usability rating: System Usability Rating Scale (SUS), Credibility and Expectancy Questionnaire (CEQ) and Intrinsic Motivation (Intrinsic Motivation). (Intrinsic Motivation Inventory, IMI) of the virtual reality application.

A.4. Subsequent evaluation: The participant's motor skills were evaluated after the three pedalling sessions, based on the pedalling sessions, based on the application of physical assessment metrics carried out by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Must had been prescribed pedalling exercise as treatment for lower limb rehabilitation caused by stroke, traumatic brain injury, neuro-motor disorders, and neuro-degenerative diseases.
* Must be able to perform a pedalling session with virtual reality technology.

Exclusion Criteria:

* An insufficient cognitive state, in particular, presence of dementia or mild cognitive impairment.
* An unbound bone fracture.
* Severe disorders of vision and/or audition (inability to perceive visual and/or auditory information coming from virtual reality)
* Those whose clinical record ruled out any incompatibility with the use of a virtual reality system.

Ages: 39 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty participants met these criteria (15 males and 5 females, mean aged=61.10, SD=12.62) diagnosed with (6) ischemic strokes, (1) hemorrhagic stroke, (1) thalamic stroke, (1) internal capsule stroke (3) traumatic brain injury (TBI), (1) Parkinson syndrome, (1) mixed axonal neuropathy with sensory demyelination, (1) progressive multifocal leukoencephalopathy, (1) secondary obstructive hydrocephalus, (1) angioma avernosus hemorrhage, (1) hemiprotuberancial hemorrhage - cavernoma, (1) ataxia and (1) cerebral artery aneurysm.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Usability of the platform | through study completion, an average of 1 month.
  Outcome of the SUS questionnaire. The score ranges from 0 to 100. A score of 72.5 or higher is considered good and above 85.0 is excellent.
Credibility and Expectancy of the platform | through study completion, an average of 1 month.
  Outcome of the CEQ questionnaire. The score ranges from 0 to 27. A score of 13.5 is considered neutral, everything above 13.5 is positive while everything under 13.5 is considered negative.
Intrinsic Motivation of the platform | through study completion, an average of 1 month.
  Outcome of the IMI questionnaire. The score ranges from 0 to 7. A score of 3.5 is considered neutral, everything above 3.5 is positive while everything under 3.5 is considered negative.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rojo, PhD Student, Study Chair — Werium Assistive Solutions
Locations (1):
- Werium Assistive Solutions, Arganda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] J. Brooke. SUS - A quick and dirty usability scale. Usability Eval. Ind., 1996; 189 (194), pp. 4-7.
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Ryan RM. Control and information in the intrapersonal sphere: an extensión of cognitive evaluation theory. J Pers Soc Psychol. 1982; 43:450-61
- [Background] Knippenberg E, Timmermans A, Palmaers S, Spooren A. Use of a technology-based system to motivate older adults in performing physical activity: a feasibility study. BMC Geriatr. 2021 Jan 28;21(1):81. doi: 10.1186/s12877-021-02021-3. PMID 33509098
- [Background] Costa V, Ramirez O, Otero A, Munoz-Garcia D, Uribarri S, Raya R. Validity and reliability of inertial sensors for elbow and wrist range of motion assessment. PeerJ. 2020 Aug 11;8:e9687. doi: 10.7717/peerj.9687. eCollection 2020. PMID 32864213
- [Background] Raya R, Garcia-Carmona R, Sanchez C, Urendes E, Ramirez O, Martin A, Otero A. An Inexpensive and Easy to Use Cervical Range of Motion Measurement Solution Using Inertial Sensors. Sensors (Basel). 2018 Aug 7;18(8):2582. doi: 10.3390/s18082582. PMID 30087258
- [Derived] Rojo A, Castrillo A, Lopez C, Perea L, Alnajjar F, Moreno JC, Raya R. PedaleoVR: Usability study of a virtual reality application for cycling exercise in patients with lower limb disorders and elderly people. PLoS One. 2023 Feb 22;18(2):e0280743. doi: 10.1371/journal.pone.0280743. eCollection 2023. PMID 36812248